CLINICAL TRIAL: NCT00898495
Title: Single Nucleotide Polymorphisms (SNP) in Platinum-/Radiation Pathway Genes to Predict Outcome in Patients With Esophageal Adenocarcinoma Treated With Cisplatin-Based Chemoradiotherapy Followed by Surgical Resection
Brief Title: Genes in Predicting Outcome in Patients With Esophageal Cancer Treated With Cisplatin, Radiation Therapy, and Surgery
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000551712; E1201T1; ASCO Foundation (Other Grant/Funding Number: ASCO)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; stage I esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Residuals from analysis

INTERVENTIONS:
Genetic: loss of heterozygosity analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict a patient's response to treatment.

PURPOSE: This laboratory study is looking at genes to see if they can predict outcome in patients with esophageal cancer treated with cisplatin, radiation therapy, and surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate patient outcomes with neoplastic cell genotypes, specifically 18 single nucleotide polymorphisms (SNPs) in 16 major genes involved in platinum metabolism and disposition and DNA repair, in patients with esophageal cancer treated with neoadjuvant cisplatin-based chemoradiotherapy followed by surgical resection on clinical trial ECOG-1201.
* Correlate patient outcomes with neoplastic cell genotypes, specifically loss of heterozygosity, in these patients.
* Correlate patient outcomes with normal (germline) cell genotypes, specifically SNPs related to platinum metabolism and disposition and DNA repair.
* Compare the predictive ability of neoplastic vs germline cell genotypes.

OUTLINE: This is a retrospective, cohort, multicenter study.

Neoplastic and normal (germline) cells are collected from pretreatment and post-treatment specimens using laser-capture microdissection. Single nucleotide polymorphisms are examined by real-time PCR. Loss of heterozygosity is assessed by analyzing short tandem repeat markers in neoplastic and germline tissue.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the esophagus

  * Stage I-IV disease
* Received cisplatin-based treatment on clinical trial ECOG-1201

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E1201
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2007-05-11 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of pretreatment clinical tumor staging vs post-treatment pathologic staging (at resection) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Harry H. Yoon, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins

REFERENCES:
- See also: Manuscript — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3118194/